CLINICAL TRIAL: NCT06402123
Title: Phase 2b Randomized, Double-blind, Placebo-controlled Crossover Study Evaluating the Efficacy and Safety of Zagociguat in Participants With MELAS (PRIZM)
Brief Title: A Phase 2b Study of Zagociguat in Patients With MELAS
Acronym: PRIZM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tisento Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIS6463-203
Record Dates: First submitted 2024-05-02; First posted 2024-05-07 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Mitochondrial Encephalopathy, Lactic Acidosis and Stroke-Like Episodes (MELAS Syndrome)
Keywords: MELAS
MeSH Terms: conditions — Mitochondrial encephalopathy; Acidosis, Lactic; MELAS Syndrome

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, 3-treatment, 2-period, incomplete-block, 4-sequence, crossover study.
  Eligible patients will be randomized to 1 of 4 crossover treatment sequences. Each treatment period will last 12 weeks, separated by a 4-week washout period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This a double-blind study in which investigators, participants/caregivers, Sponsor, and all study personnel will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo then Zagociguat 15mg (Experimental): Participants first receive placebo once a day for 12 weeks. Then after a 4 week washout, they receive zagociguat 15 mg once a day for 12 weeks.
  Interventions: Drug: zagociguat 15mg; Drug: Placebo
- Zagociguat 15mg then Placebo (Experimental): Participants first receive zagociguat 15 mg once a day for 12 weeks. Then after a 4-week washout, they receive placebo once a day for 12 weeks.
  Interventions: Drug: zagociguat 15mg; Drug: Placebo
- Placebo then Zagociguat 30mg (Experimental): Participants first receive placebo once a day for 12 weeks. Then after a 4-week washout, they receive zagociguat 30 mg once a day for 12 weeks.
  Interventions: Drug: zagociguat 30mg; Drug: Placebo
- Zagociguat 30mg then Placebo (Experimental): Participants first receive zagociguat 30 mg once a day for 12 weeks. Then after a 4-week washout, they receive placebo once a day for 12 weeks.
  Interventions: Drug: zagociguat 30mg; Drug: Placebo

INTERVENTIONS:
Drug: zagociguat 15mg — Once-daily oral tablets
  Other Names: IW-6463; CY6463
  Arms: Placebo then Zagociguat 15mg; Zagociguat 15mg then Placebo
Drug: zagociguat 30mg — Once-daily oral tablets
  Other Names: IW-6463; CY6463
  Arms: Placebo then Zagociguat 30mg; Zagociguat 30mg then Placebo
Drug: Placebo — Once-daily oral tablets

SUMMARY:
PRIZM is a Phase 2b randomized, double-blind, placebo-controlled, 3-treatment, 2-period, crossover study evaluating the efficacy and safety of oral zagociguat 15 and 30 mg vs. placebo when administered daily for 12 weeks in participants with genetically and phenotypically defined MELAS.

DETAILED DESCRIPTION:
The goal of this clinical trial is to learn about the effectiveness of zagociguat in patients with MELAS. The main questions it aims to answer are:

* Does zagociguat improve fatigue in patients with MELAS?
* Does zagociguat improve cognitive performance in patients with MELAS?
* What is the safety and tolerability profile of zagociguat?

The PRIZM study is evaluating 2 dose levels of zagociguat in a crossover design consisting of two 12-week treatment periods separated by a 4-week washout. Patients will be screened and if eligible, randomly assigned either to receive placebo in period 1 followed by active drug in period 2 OR to receive active drug in period 1 followed by placebo in period 2. Study medication is a once daily oral tablet and will be provided at the clinic and/or shipped to the participant's home. Clinic visits will occur at screening and Week 1 and Week 12 of each treatment period. Visits at Week 4 and Week 8 of both crossover periods will either be in clinic or optionally at the participant's home. Study assessments will be conducted weekly on a phone app and a separate tablet and additional assessments will be conducted during visits. Patients who complete the study will be eligible for an open label extension study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent form.
2. 18 to 75 years of age.
3. Diagnosed with MELAS based on the presence of each of the following criteria:

   1. A documented pathogenic variant in a mitochondrial DNA (mtDNA) gene.
   2. History of one or more stroke-like episodes (SLEs) with magnetic resonance imaging (MRI) findings consistent with stroke-like lesions.
4. Scores below normal average on the iDSST and GMLT.
5. Reports fatigue due to MELAS.
6. Can complete at least 1 sit-to-stand in the 30-second test interval.
7. Completes all at-home weekly activities independently during the Screening Period (caregiver may help set up device/app, log-in, etc.).
8. Other criteria per the protocol.

Exclusion Criteria:

1. Systolic blood pressure (BP) 90 mmHg or diastolic BP 60 mmHg.
2. Orthostatic hypotension when measured after standing from a semi-recumbent/supine position.
3. Active cancer significant enough to confound the results of this study.
4. Severe gastrointestinal dysmotility that may impact participation.
5. Recent history (within last 6 months) of platelet dysfunction, hemophilia, von Willebrand disease, coagulation disorder, other bleeding diathesis condition(s), or significant, nontraumatic bleeding episodes.
6. History of spontaneous fracture(s) that in the investigator's opinion represents a safety risk for trial participation.
7. Current use of prohibited medication (reviewed by investigator).
8. Any medical or other condition that the investigator thinks would preclude study participation.
9. Other exclusion criteria per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
• PROMIS Fatigue MELAS Short Form scores• Groton Maze Learning Test scores • International Digit Symbol Substitution Test scores | Weeks 9 through 12 of each treatment period
  These measures are a patient reported questionnaire on MELAS-specific fatigue and 2 cognitive performance tests. These 3 outcome measures will be combined using a global statistical test.
Incidence of Treatment-emergent Adverse Events (TEAEs) | Weeks 1 through washout for treatment period 1 and Weeks 1 through follow-up for treatment period 2
  TEAEs are any untoward event that may or may not be related to study medication.

SECONDARY OUTCOMES:
Number of repetitions completed during the 30-second sit-to-stand test | Week 12
  Leg strength and exercise intolerance
PROMIS Cognitive Function MELAS Short Form (PCFM-SF) score | Week 12
  Patient-reported questionnaire on MELAS-specific cognitive function
Plasma concentrations of GDF-15 | Week 12
  Measure of disease pathophysiology
Memory composite scores (One Card Learning and One Back Tests) for Week 9 through 12 | Week 9 through 12
  Test of memory

CONTACTS AND LOCATIONS:
Locations (21):
- United States (11):
  - UC San Diego - Altman Clinical and Translational Research Institute, La Jolla, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Rare Disease Research, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Mount Sinai - Ichan School of Medicine, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Medical School at Houston, Houston, Texas
- Australia (2):
  - Neuroscience Research Australia, Sydney, New South Wales
  - Royal Melbourne Hospital, Melbourne, Victoria
- Canada (2):
  - Shared Health/University of Manitoba, Winnipeg, Manitoba
  - McMaster University Medical Center, Hamilton, Ontario
- Germany (2):
  - University Hospital Bonn, Bonn
  - Ludwig-Maximilians-University of Munich, Munich
- Italy (2):
  - Neurologic Institute Carlo Besta of Milan, Milan
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- United Kingdom (2):
  - UCL Queen Square Institute of Neurology, London
  - Newcastle University, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No